CLINICAL TRIAL: NCT04562181
Title: Consistency Evaluation of the qCON, qNOX Indices and Bispectral Index in Detecting Hypnotic and Nociception Level During and After General Anesthesia in Gastrointestinal Surgery Patients
Brief Title: Consistency Evaluation of the qCON, qNOX Indices and Bispectral Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20200915
Record Dates: First submitted 2020-09-14; First posted 2020-09-24 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Anesthesia Monitor; Electroencephalography; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventions (Experimental): Anesthesia will be induced with bolus infusion using propofol, sufentanil and cis-atracurium intravenously. The patients will be intubated subsequently. TOF (T4/T1) will be calculated continuously using muscle relaxation monitoring. Anesthesia are maintained with a combination of sevoflurane, propofol, sufentanil and cis-atracurium. Anti-emetic and opioids will be routinely administrated prior to abdominal closure. Neostigmine will be administrated for reversing the residual neuromuscular blockade after the patient get his breath. Tracheal extubating is indicated by a TOF value above 70% in addition to other physical signs.
  Interventions: Other: Bispectral index and qCON/qNOX monitoring

INTERVENTIONS:
Other: Bispectral index and qCON/qNOX monitoring — This study will characterise the bispectral index data and qCON/qNOX index data in 30 patients during the operation and first postoperative night

SUMMARY:
The first objective of this work is to compare the performances of three electroencephalogram based indices, the qCON index, the qNOX index and the bispectral index (BIS), in patients receiving gastrointestinal surgery during first postoperative night. Secondly, their behaviors under general anesthesia are also pointed out.

The qCON and qNOX indices are implemented in an Angel 6000 monitor (WellHealth Medical Co Ltd., Shenzhen, China), and BIS indices are recorded in a BIS monitor (Aspect Medical Systems, Norwood, MA, USA).

Data will be obtained from 30 patients scheduled for selective surgery undergoing general anesthesia with a combination of propofol, sufentanil and cis-atracurium in the first Hospital of China Medical University. The values of qCON, qNOX and BIS were statistically compared. The qCON, qNOX indices are recorded together with BIS during the whole operation period (Awake- Anesthesia-Recovery stages), as well as during the first night postoperatively (from 8:00pm to 06:00am). The values of qCON, qNOX and BIS were statistically compared. The Consistency evaluation will be conducted between qCON/qNOX and BIS.

DETAILED DESCRIPTION:
This study was approved by the ethics committee of China Medical University. The study will be carried out in the 1st Hospital of China Medical University. Thirty patients scheduled for selective gastrointestinal surgery undergoing general anesthesia will be enrolled. There are two steps in this study: In step1, The qCON and qNOX indices will be continuously recorded throughout the whole surgery, using a Angel-6000 monitor (WellHealth Medical Co Ltd., Shenzhen, China). Meanwhile, the bispectral index (BIS) will be recorded using Aspect BIS monitor (Aspect Medical Systems, Norwood, MA, USA) in the same patient in order to compare with qCON and qNOX.

The general anesthesia protocol is as following: Anesthesia will be induced with bolus infusion of propofol, sufentanil and cis-atracurium intravenously. The patients will be intubated subsequently. TOF (T4/T1) value will be observed throughout using muscle relaxation monitoring (GE healthcare, USA). Anesthesia are maintained with a combination of sevoflurane, propofol, sufentanil and cis-atracurium. Dosage of the anesthetics will be adjusted according to the BIS value and hemodynamics fluctuating. Anti-emetic and opioids will be routinely administrated prior to abdominal closure. Neostigmine will be administrated for reversing the residual neuromuscular blockade after the patient get his breath. Tracheal extubating is indicated by a TOF value above 70% in addition to other physical signs. The qCON, qNOX and BIS indices will be continuously recorded before anesthesia induction (fully awake), during the operation (sleep) and after the operation (fully recovery). The dosage of propofol, sufentanil and cis-atracurium used in the operation are also recorded.

In step2, all these three electroencephalogram-based indices are collected again at the 1st postoperative night. The Angel-6000 and Aspect BIS monitor will be placed again to the identical patient who have received the operation on the daytime. Data collecting period is from 8:00 pm to 6:00 am the next day. Sleep was defined as the duration of BIS value below 80 in the 10 hours of monitoring (from 8:00pm to 6:00am).

If there are specific requirements for management with regards to postoperative pain or any other anesthesia related complications, name and the dosage of the treatments will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese;
* Age: from 18 to 80 years old;
* Hospitalized patients

Exclusion Criteria:

* Cognitive difficulties
* Mental diseases
* Without an informed consent
* Inability to cooperate with the researcher's requirements
* Deprivation of the human right by an administrative or juridical entity
* Ongoing participation or participation in another study within 1 month
* Night surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
qCON/qNOX indices of the first postoperative night | on the first postoperative night
  This study will characterise the qCON/qNOX index data in 30 patients during first postoperative night

SECONDARY OUTCOMES:
qCON/qNOX indices data during operation | from the beginning to the end of surgery
  This study will characterise qCON/qNOX index data in 30 patients receiving gastrointestinal surgery under general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Wen-fei Tan, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided